CLINICAL TRIAL: NCT07005167
Title: Clinical Performance of Endocrowns Fabricated From Two Hybrid Ceramic Materials on Endodontically Treated Molars: A Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Ahmed Farid Zaki Shehab, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 240789; Shofu Inc, (Other: Shofu Japan)
Record Dates: First submitted 2025-06-03; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Endocrown Restoration
Keywords: Hybrid ceramics; cerasmart; HC hard blocks

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double-blind clinical trial with 1:1 allocation ratio.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatients with endo-treated molars that will be restored with HC hard hybrid ceramic endocrowns (Experimental)
  Interventions: Procedure: endocrowns
- utpatients with endo-treated molars that will be restored with Cerasmart endocrowns (Active Comparator)
  Interventions: Procedure: endocrowns

INTERVENTIONS:
Procedure: endocrowns — endocrowns made of HC hard blocks or cerasmart blocks to restore endo treated molars
  Arms: Outpatients with endo-treated molars that will be restored with HC hard hybrid ceramic endocrowns
Procedure: endocrowns — endocrowns made of Cerasmart blocks to restore endo treated molars
  Arms: utpatients with endo-treated molars that will be restored with Cerasmart endocrowns

SUMMARY:
The goal of this study is to evaluate the clinical success rate (measured by retention) of endo-crowns fabricated from two hybrid ceramic materials (HC Hard blocks ) versus (Cerasmart) at 6, 12, and 18 months.

Secondary Objectives are:

1. To compare the incidence of restoration failures between the two materials
2. To assess marginal adaptation and marginal discoloration over time
3. To evaluate wear of opposing enamel quantitatively
4. To compare surface texture, color match, and luster between materials
5. To determine patient satisfaction with both types of restorations It will be a randomized, controlled, double-blind clinical trial with 1:1 allocation ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥21 years
2. Good general health (ASA I or II)
3. Willing and able to provide informed consent
4. Committed to follow-up appointments for 18 months
5. Root canal treated molars requiring restoration
6. Adequate remaining tooth structure:

   * Minimum 2mm ferrule height
   * Sufficient wall thickness (≥1.5mm)
   * At least 2 remaining walls
7. Opposing natural dentition or fixed prosthesis
8. Adequate periodontal health:

   * Probing depth ≤4mm
   * No bleeding on probing
9. Good oral hygiene with plaque score ≤20%
10. Sufficient mouth opening for clinical procedures
11. Normal occlusion and acceptable interocclusal space

Exclusion Criteria:

1. Pregnant or lactating women
2. Severe bruxism or parafunctional habits
3. Active periodontal disease
4. Active caries or inadequate oral hygiene
5. Less than 2mm ferrule height after preparation
6. Apical pathology or inadequate root canal treatment
7. Tooth mobility grade II or III
8. Known allergy to materials used
9. Uncontrolled diabetes (HbA1c >7.0%)
10. Radiation therapy in head and neck region
11. Temporomandibular joint disorders
12. History of poor compliance with dental appointments
13. Heavy smokers (>10 cigarettes/day)
14. Chronic use of medications affecting salivary flow
15. Unable to understand study requirements
16. Evidence of pulpal or periapical pathology

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Retention | From cementation of endocrown, then at 6 months, 12 months and 18 months
  Modified USPHS criteria

SECONDARY OUTCOMES:
Restoration Failure | From cementation of endocrown, then at 6 months, 12 months and 18 months
  Modified USPHS criteria
Marginal Adaptation | From cementation of endocrown, then at 6 months, 12 months and 18 months
  Modified USPHS criteria
Wear of Opposing Enamel | From cementation of endocrown, then at 6 months, 12 months and 18 months
  Digital software (Geomagic)
Surface Texture | From cementation of endocrown, then at 6 months, 12 months and 18 months
  Modified USPHS criteria
Color Match | From cementation of endocrown, then at 6 months, 12 months and 18 months
  Modified USPHS criteria
Luster of Restoration | From cementation, then at 6 months, 12 months and 18 months
  Modified USPHS criteria
Patient Satisfaction | From cementation, then at 6 months, 12 months and 18 months
  VAS (Questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided